CLINICAL TRIAL: NCT05149235
Title: Effects of Infusion of Gaming Technology With Cardiac Rehabilitation on Autonomic Modulation of Heart: a Randomized Control Trial
Brief Title: Gaming Technology and Cardiac Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahria University (Other)
Responsible Party: Principal Investigator, Seyyada Tahniat Ali, clinical instructor, Bahria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FRC-BUMDC 23/2021
Record Dates: First submitted 2021-11-02; First posted 2021-12-08 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Open Heart Surgery
Keywords: Cardiac rehabilitation; autonomic regulation of heart; physical activity; gaming technology; cycle ergometer
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- early mobilization group (Active Comparator): this group will perform early mobilization exercises using a cycle ergometer.
  Interventions: Other: early mobilization group
- game tech group (Experimental): this group will use physio adventure device instead of a cycle ergometer
  Interventions: Device: physio adventure
- placebo group (Placebo Comparator): this group is placebo control and will receive routine respiratory physiotherapy
  Interventions: Other: placebo

INTERVENTIONS:
Other: early mobilization group — Participants will perform exercises using only the cycle ergometer and ambulation. In this group, participants will be instructed to turn the pedals continuously, without any weight added to the equipment (only on 1st post-operative day) and training load will be determined by a fatigue level maintenance of 4 or 5 on the modified Borg scale with a maximum HR elevation of 20% on 2nd and 3rd post-operative days. Duration of exercise will be of 10 minutes (five minutes with the upper limbs and five minutes with the lower limbs). For the arm exercises, the individuals will be positioned with the head end of the bed raised to 60° above the horizontal, while ensuring that all the equipment responsible for measuring the patient's vital signs remained connected. For the leg exercises, the head end of the bed will be lowered to a 30° angle to provide better access to the pedals and avoid compensatory hip movements. Ambulation will be performed only on 3rd post-operative day (40 meters).
  Arms: early mobilization group
Device: physio adventure — The protocol applied to the experimental group will be the same of that applied to the early mobilization group with the use of smart move instead of cycle ergometer.
  Arms: game tech group
Other: placebo — Participants allocated to the Control group will perform respiratory physiotherapy (Flow-oriented incentive spirometer (3×15), active exercises for lower and upper limbs, with each movement being repeated 10 times in an open kinetic chain. For the upper limbs, movements of anterior flexion of the shoulder will be performed until achieving maximum range of motion, using diagonal movements starting at the contralateral iliac crest up to the maximum range of anterior flexion of the shoulder associated with supination. For the lower limbs, exercises will consist of straight leg raises, hip and knee flexion-extension exercise and ankle pumps. Sessions will be of 10 minutes duration.
  Arms: placebo group

SUMMARY:
Moderate to vigorous physical activity has been shown to be associated with autonomic regulation of the heart measured with heart rate variability. Cardiac autonomic modulation can be evaluated by heart rate variability. Activity promoting games can be an effective tool to aid rehabilitation in clinical settings. Combining gaming with the ergo-cycle can facilitate improving patients' activity time spent on the cycle.

DETAILED DESCRIPTION:
Physical activity is recognized as a central component of cardiac rehabilitation, improving control of cardiovascular risk factors, reducing the incidence of adverse events, leading to improvements in cardiovascular conditioning and prevention of thromboembolic events. Consequently, it provides greater physical independence and safety for hospital discharge. Coronary artery bypass grafting (CABG) surgery may lead to prolonged bed rest, and immobility, which can result in negative consequences, such as a decrease in functional capacity, decrease in muscle mass and muscle tone, postural hypotension, and changes in autonomic modulation of the heart rate. Cardiac autonomic modulation can be evaluated by heart rate variability (HRV), which involves simple noninvasive measurement of the oscillations in intervals between consecutive heartbeats.

Technology such as video games plays a complicated role in physical inactivity-much like a double-edged sword. To overcome this problem, the newly emerged active video games have been increasingly used to promote physical activity and health among various populations. Augmented reality games are unique because they integrate the physical and virtual worlds into a single interface using mobile devices applications. Investigators present a proof of concept of an endless running game called physio adventure which implements an activity recognition system that detects cycle rotation and its speed. The goal is to replace the traditional rehabilitation devices with innovative gaming technology with a more natural movement-based one, showing the potential of this kind of interaction to create innovative and immersive experiences while promoting physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to elective cardiac surgery (valvular or coronary bypass surgery by sternotomy)
* Both male and female
* a score of 15 on the Glasgow Coma Scale
* musculoskeletal, and cardiopulmonary conditions suitable for the accomplishment of the proposed activities
* absence of neurological sequelae and/or neurodegenerative diseases

Exclusion Criteria:

* Those who had difficulty understanding the activities involved in the study.
* those with any motor or neurological impairment that would prevent them from using a cycle ergometer.
* those who discontinued the protocol on the ward for return to the ICU
* previous cardiac surgeries
* hemodynamic instability that prevented protocol performance
* breathing discomfort
* invasive ventilatory support
* oxygen saturation below 90% (even with complementary oxygen therapy)
* coagulation disorders
* infections in any of the systems
* nonperformance of the whole protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
change in autonomic modulation of heart | heart rate variability will be recorded on day of admission, 1st post-operative day and 4th post operative day
  autonomic modulation of heart will be assessed by measuring heart rate variability

CONTACTS AND LOCATIONS:
Overall Officials: Seyyada T Ali, Principal Investigator — bahria university medical and dental college; muhammad i tariq, Study Director — Riphah International University; urooj fatima, Study Chair — bahria university medical and dental college
Locations (1):
- Seyyada Tahniat Ali, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] European Association of Cardiovascular Prevention and Rehabilitation Committee for Science Guidelines; EACPR; Corra U, Piepoli MF, Carre F, Heuschmann P, Hoffmann U, Verschuren M, Halcox J; Document Reviewers; Giannuzzi P, Saner H, Wood D, Piepoli MF, Corra U, Benzer W, Bjarnason-Wehrens B, Dendale P, Gaita D, McGee H, Mendes M, Niebauer J, Zwisler AD, Schmid JP. Secondary prevention through cardiac rehabilitation: physical activity counselling and exercise training: key components of the position paper from the Cardiac Rehabilitation Section of the European Association of Cardiovascular Prevention and Rehabilitation. Eur Heart J. 2010 Aug;31(16):1967-74. doi: 10.1093/eurheartj/ehq236. Epub 2010 Jul 19. PMID 20643803
- [Background] Gama Lordello GG, Goncalves Gama GG, Lago Rosier G, Viana PADC, Correia LC, Fonteles Ritt LE. Effects of cycle ergometer use in early mobilization following cardiac surgery: a randomized controlled trial. Clin Rehabil. 2020 Apr;34(4):450-459. doi: 10.1177/0269215520901763. Epub 2020 Jan 29. PMID 31994405
- [Background] Cacau Lde A, Oliveira GU, Maynard LG, Araujo Filho AA, Silva WM Jr, Cerqueria Neto ML, Antoniolli AR, Santana-Filho VJ. The use of the virtual reality as intervention tool in the postoperative of cardiac surgery. Rev Bras Cir Cardiovasc. 2013 Jun;28(2):281-9. doi: 10.5935/1678-9741.20130039. PMID 23939326
- [Background] Kulur AB, Haleagrahara N, Adhikary P, Jeganathan PS. Effect of diaphragmatic breathing on heart rate variability in ischemic heart disease with diabetes. Arq Bras Cardiol. 2009 Jun;92(6):423-9, 440-7, 457-63. doi: 10.1590/s0066-782x2009000600008. English, Multiple languages. PMID 19629309
- [Background] Karapolat H, Engin C, Eroglu M, Yagdi T, Zoghi M, Nalbantgil S, Durmaz B, Kirazli Y, Ozbaran M. Efficacy of the cardiac rehabilitation program in patients with end-stage heart failure, heart transplant patients, and left ventricular assist device recipients. Transplant Proc. 2013 Nov;45(9):3381-5. doi: 10.1016/j.transproceed.2013.06.009. PMID 24182820
- [Background] Oliveira NL, Ribeiro F, Alves AJ, Teixeira M, Miranda F, Oliveira J. Heart rate variability in myocardial infarction patients: effects of exercise training. Rev Port Cardiol. 2013 Sep;32(9):687-700. doi: 10.1016/j.repc.2013.02.010. Epub 2013 Aug 30. PMID 23993292
- [Background] Gao Z. Fight fire with fire? Promoting physical activity and health through active video games. J Sport Health Sci. 2017 Mar;6(1):1-3. doi: 10.1016/j.jshs.2016.11.009. Epub 2016 Nov 24. No abstract available. PMID 30356540
- [Background] Baranowski T. Pokemon Go, go, go, gone? Games Health J. 2016 Oct;5(5):293-294. doi: 10.1089/g4h.2016.01055.tbp. Epub 2016 Aug 15. No abstract available. PMID 27525347
- [Background] Pasco D, Roure C, Kermarrec G, Pope Z, Gao Z. The effects of a bike active video game on players' physical activity and motivation. J Sport Health Sci. 2017 Mar;6(1):25-32. doi: 10.1016/j.jshs.2016.11.007. Epub 2016 Nov 24. PMID 30356595
- [Background] Ribeiro BC, Poca JJGD, Rocha AMC, Cunha CNSD, Cunha KDC, Falcao LFM, Torres DDC, Rocha LSO, Rocha RSB. Different physiotherapy protocols after coronary artery bypass graft surgery: A randomized controlled trial. Physiother Res Int. 2021 Jan;26(1):e1882. doi: 10.1002/pri.1882. Epub 2020 Oct 25. PMID 33103326